CLINICAL TRIAL: NCT02691533
Title: To Study the Immunomodulating Effects and Safety Profile of ω3 and ω6 PUFA Containing Intravenous Lipid Emulsion in Patients With Acute on Chronic Liver Failure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institute of Liver and Biliary Sciences, India (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ILBS-ACLF-006
Record Dates: First submitted 2016-02-15; First posted 2016-02-25 (Estimated); Last update posted 2018-09-05 (Actual); Status verified 2018-02

CONDITIONS: Chronic Liver Failure
Keywords: Acute
MeSH Terms: conditions — End Stage Liver Disease | interventions — Fatty Acids, Unsaturated; soybean oil, phospholipid emulsion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- ω3 PUFA(10% Omegavan 100 ml) (Experimental)
  Interventions: Drug: ω3 PUFA (Polyunsaturated fatty acids) (10% Omegavan 100 ml)
- ω6 PUFA (20% Intralipid 50 ml) (Experimental)
  Interventions: Drug: ω6 PUFA (Polyunsaturated fatty acids) (10% Intralipid 100 ml)
- Placebo Arm (Placebo Comparator): No Lipid Emulsion will be given in this arm
  Interventions: Drug: No Lipid Emulsion/Placebo

INTERVENTIONS:
Drug: ω3 PUFA (Polyunsaturated fatty acids) (10% Omegavan 100 ml)
  Arms: ω3 PUFA(10% Omegavan 100 ml)
Drug: ω6 PUFA (Polyunsaturated fatty acids) (10% Intralipid 100 ml)
  Arms: ω6 PUFA (20% Intralipid 50 ml)
Drug: No Lipid Emulsion/Placebo
  Arms: Placebo Arm

SUMMARY:
Study population: Patients admitted or seen in OPD (Out Patient Department), Department of Hepatology.

Study design- Prospective Randomized Controlled Trial. Study period-January 2016 to May 2017 Intervention- Subjects will be randomized into 3 groups Group A subjects will receive ω3 PUFA (Polyunsaturated Fatty Acids) (10% Omegavan 100 ml).

Group B- will receive ω6 PUFA (Polyunsaturated Fatty Acids) (10% Intralipid 100 ml).

Group C -Placebo group

Monitoring and assessment- :- The following tests will be done in these patients:-

1. Complete clinical examination.
2. Serum electrolytes- sodium, potassium, calcium, magnesium, phosphate levels
3. BUN (Blood Urea Nitrogen)
4. Serum free fatty acid levels
5. Lipid profile.
6. Arterial ammonia
7. Arterial lactate
8. Blood sugar and serum insulin levels

ELIGIBILITY:
Inclusion Criteria:

* Acute on Chronic Liver Failure (ACLF) patients aged 18 years and above
* Patients tolerating enteral nutrition
* Patients with no overt sepsis - no fever, sterile blood and urine cultures, procalcitonin <2

Exclusion Criteria:

* Active ongoing GI bleed
* Allergy to soya oil, eggs, peanuts or other ingredients of intralipid.
* Co-morbidities like Diabetes mellitus, hyperlipidemia, CAD and hypothyroidism.
* Renal failure (S.creatinine > 2.5mg%)
* Pregnancy
* Patients with shock requiring vasopressor support
* Patients on anticoagulants
* Refusal to participate in the study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2016-02-01 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
Effect of intravenous lipid emulsions (w3/ w6) on systemic inflammation and endotoxemia levels at the end of 5 days. | 5 days
  Decrease in endotoxins levels , TNF alpha,ilnterleukin 6,ilnterleukin 10,Monocyte/ macrophage activation etc.
  All of them are markers of inflammation. The outcome systemic inflammation is a composite outcome which includes all the above mentioned markers

SECONDARY OUTCOMES:
Incidence of sepsis and related complications | 28 days
Effect of lipid infusion (w3/w6) on metabolic parameters viz., serum triglyceride levels, serum ketone levels, free fatty acid levels and arterial lactate levels. | 5 days
  Metabolic parameter is a composite outcome of all the above said markers.
Influence of lipid infusion (w3/w6) on nitrogen balance. | 5 days
  Improvement or deterioration in urinary urea nitrogen.
Effect of lipid infusion (w3/w6) on International Normalized Ratio (INR). | 5 days
  Effect is defined as INR (International Normalized Ratio) value within normal limit or improvement as compare to baseline value.
Oxidative stress response to lipid infusion | 5 days
  Oxidative stress response is based on the Improvement or deterioration in Isoprostane levels in urine
Influence of lipid infusion(w3/w6) on 28day mortality | 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Dr Anand Kulkarni V, MD, Principal Investigator — Institute of Liver and Biliary Sciences
Locations (1):
- Institute of liver and Biliary Sciences, New Delhi, National Capital Territory of Delhi, India

IPD SHARING:
Plan to Share IPD: No